CLINICAL TRIAL: NCT00673790
Title: Blood Pressure and Metabolic Effects of Nebivolol Compared With Hydrochlorothiazide and Placebo in Hypertensive Patients With Impaired Glucose Tolerance or Impaired Fasting Glucose
Brief Title: The Blood Pressure and Metabolic Effects of Nebivolol in Hypertensive Patients With Impaired Glucose Tolerance or Impaired Fasting Glucose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB-MD-04
Record Dates: First submitted 2008-04-29; First posted 2008-05-07 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Hypertension
Keywords: nebivolol; BYSTOLIC ™; hydrochlorothiazide; lisinopril; Prinivil (TM); Zestril (TM); losartan; Cozaar (TM); Impaired Fasting Glucose; Impaired Glucose Tolerance; hypertension
MeSH Terms: conditions — Hypertension; Glucose Intolerance | interventions — Nebivolol; Lisinopril; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nebivolol (Active Comparator): Nebivolol with concomitant losartan or lisinopril
  Interventions: Drug: Nebivolol with concomitant losartan or lisinopril
- Hydrochlorothiazide (HCTZ) (Active Comparator): HCTZ with concomitant losartan or lisinopril
  Interventions: Drug: HCTZ with concomitant losartan or lisinopril
- Placebo (Placebo Comparator): Placebo with concomitant losartan or lisinopril
  Interventions: Drug: Placebo with concomitant losartan or lisinopril

INTERVENTIONS:
Drug: Nebivolol with concomitant losartan or lisinopril — Encapsulated Nebivolol 5 mg, 10 mg, 20, mg, 40 mg total daily dosage, oral administration with concomitant treatment consisting of lisinopril 10 mg total daily dosage, oral administration or losartan 50 mg total daily dosage, oral administration.
  Arms: Nebivolol
Drug: HCTZ with concomitant losartan or lisinopril — Encapsulated Hydrochlorothiazide 12.5 mg or 25 mg total daily dosage, oral administration with concomitant treatment consisting of lisinopril 10 mg total daily dosage, oral administration or losartan 50 mg total daily dosage, oral administration.
  Arms: Hydrochlorothiazide (HCTZ)
Drug: Placebo with concomitant losartan or lisinopril — Placebo with concomitant treatment consisting of lisinopril 10 mg total daily dosage, oral administration or losartan 50 mg total daily dosage, oral administration.
  Arms: Placebo

SUMMARY:
This study is being done to see if the blood pressure and metabolic effects of an approved drug nebivolol is comparable to that of another approved drug hydrochlorothiazide (HCTZ) and placebo in hypertensive patients.

DETAILED DESCRIPTION:
This study is double blind (neither you nor the physician will know when you are receiving placebo, which is an inactive compound such as a sugar pill, or active study drugs nebivolol or hydrochlorothiazide).

All participants will also receive lisinopril, an angiotensin converting enzyme, or losartan, an angiotensin receptor blocker. All medications are approved and marketed for the treatment of hypertension.This study is being conducted in about 500 patients at approximately 80 research centers in the United States.

The study consists of approximately 9 study visits over a period of 5 months. During these visits, patients will undergo routine health exams and some special laboratory tests such as an oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ambulatory outpatients 18-80 years old at screening.
* Have a history of hypertension and taking up to 2 medications for high blood pressure.
* Qualifying laboratory results confirming impaired fasting glucose or impaired glucose tolerance
* Vision and hearing (hearing aid permissible) sufficient for compliance with questionnaire completion

Exclusion Criteria:

* Have clinically significant respiratory, liver or cardiovascular disease
* Presence of coronary artery disease requiring treatment with a beat blocker, calcium channel blocker or nitrates
* Use of niacin or antidiabetic drugs (oral or injectable) within 6 months before study entry
* Have a history of hypersensitivity to nebivolol, other beta-blockers, hydrochlorothiazide, or other sulfonamide-derived drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2008-05-15 (Actual); Primary Completion 2010-07-09 (Actual); Study Completion 2010-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Shea, MS, Study Director — Forest Research Institute, a subdisiary of Forest Laboratories, Inc.
Locations (88):
- United States (88):
  - Forest Investigative Site 058, Athens, Alabama
  - Forest Investigative Site 101, Birmingham, Alabama
  - Forest Investigative Site 016, Huntsville, Alabama
  - Forest Investigative Site 119, Phoenix, Arizona
  - Forest Investigative Site 078, Tucson, Arizona
  - Forest Investigative Site 056, Anaheim, California
  - Forest Investigative Site 097, Bell Gardens, California
  - Forest Investigative Site 026, Buena Park, California
  - Forest Investigative Site 147, Buena Park, California
  - Forest Investigative Site 061, Chino, California
  - Forest Investigative Site 108, Costa Mesa, California
  - Forest Investigative Site 054, Encinitas, California
  - Forest Investigative Site 128, Fresno, California
  - Forest Investigative Site 127, Huntington Park, California
  - Forest Investigative Site 030, Long Beach, California
  - Forest Investigative Site 085, Los Angeles, California
  - Forest Investigative Site 028, Los Angeles, California
  - Forest Investigative Site 124, National City, California
  - Forest Investigative Site 117, Riverside, California
  - Forest Investigative Site 025, Roseville, California
  - Forest Investigative Site 017, Sacramento, California
  - Forest Investigative Site 068, San Diego, California
  - Forest Investigative Site 112, Santa Ana, California
  - Forest Investigative Site 063, Temecula, California
  - Forest Investigative Site 013, Tustin, California
  - Forest Investigative Site 052, Walnut Creek, California
  - Forest Investigative Site 074, Milford, Connecticut
  - Forest Investigative Site 139, Brooksville, Florida
  - Forest Investigative Site 103, Coral Gables, Florida
  - Forest Investigative Site 019, Daytona Beach, Florida
  - Forest Investigative Site 010, DeLand, Florida
  - Forest Investigative Site 073, Hialeah, Florida
  - Forest Investigative Site 109, Hialeah, Florida
  - Forest Investigative Site 036, Hollywood, Florida
  - Forest Investigative Site 104, Miami, Florida
  - Forest Investigative Site 121, Miami, Florida
  - Forest Investigative Site 099, Miami, Florida
  - Forest Investigative Site 107, Pembroke Pines, Florida
  - Forest Investigative Site 141, St. Petersburg, Florida
  - Forest Investigative Site 140, Tampa, Florida
  - Forest Investigative Site 060, West Palm Beach, Florida
  - Forest Investigative Site 125, West Palm Beach, Florida
  - Forest Investigative Site 075, Atlanta, Georgia
  - Forest Investigative Site 072, Atlanta, Georgia
  - Forest Investigative Site 042, Augusta, Georgia
  - Forest Investigative Site 094, Honolulu, Hawaii
  - Forest Investigative Site 95, Meridian, Idaho
  - Forest Investigative Site 082, Chicago, Illinois
  - Forest Investigative Site 096, Wichita, Kansas
  - Forest Investigative Site 065, Madisonville, Kentucky
  - Forest Investigative Site 123, Lafayette, Louisiana
  - Forest Investigative Site 106, Auburn, Maine
  - Forest Investigative Site 006, Oxon Hill, Maryland
  - Forest Investigative Site 067, Brockton, Massachusetts
  - Forest Investigative Site 110, Brockton, Massachusetts
  - Forest Investigative Site 018, Paw Paw, Michigan
  - Forest Investigative Site 021, Saint Clair Shores, Michigan
  - Forest Investigative Site 080, Columbia, Missouri
  - Forest Investigative Site 146, Elizabeth, New Jersey
  - Forest Investigative Site 071, Brooklyn, New York
  - Forest Investigative Site 081, New York, New York
  - Forest Investigative Site 035, Charlotte, North Carolina
  - Forest Investigative Site 051, Charlotte, North Carolina
  - Forest Investigative Site 077, Durham, North Carolina
  - Forest Investigative Site 100, Lenoir, North Carolina
  - Forest Investigative Site 041, Morehead City, North Carolina
  - Forest Investigative Site 050, Salisbury, North Carolina
  - Forest Investigative Site 091, Centerville, Ohio
  - Forest Investigative Site 089, Cincinnati, Ohio
  - Forest Investigative Site 122, Perrysburg, Ohio
  - Forest Investigative Site 087, Eugene, Oregon
  - Forest Investigative Site 088, Portland, Oregon
  - Forest Investigative Site 114, Harleysville, Pennsylvania
  - Forest Investigative Site 083, Pawtucket, Rhode Island
  - Forest Investigative Site 098, Columbia, South Carolina
  - Forest Investigative Site 115, Greer, South Carolina
  - Forest Investigative Site 105, Simpsonville, South Carolina
  - Forest Investigative Site 092, Sioux Falls, South Dakota
  - Forest Investigative Site 003, Carrollton, Texas
  - Forest Investigative Site 116, Houston, Texas
  - Forest Investigative Site 120, Odessa, Texas
  - Forest Investigative Site 012, San Antonio, Texas
  - Forest Investigative Site 048, Sugar Land, Texas
  - Forest Investigative Site 040, Bountiful, Utah
  - Forest Investigative Site 062, Salt Lake City, Utah
  - Forest Investigative Site 093, Salt Lake City, Utah
  - Forest Investigative Site 130, West Jordan, Utah
  - Forest Investigative Site 126, Arlington, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: May 2008 to March 2010 at 96 US sites, 72 sites randomized patients.
Pre-assignment Details: A losartan or lisinopril run-in phase was required for all patients before assignment to Placebo or Nebivolol or Hydrochlorothiazide arms.
Groups:
- Nebivolol: Encapsulated Nebivolol 5 mg, 10 mg, 20, mg, 40 mg total daily dosage, oral administration with concomitant treatment consisting of lisinopril 10 mg total daily dosage, oral administration or losartan 50 mg total daily dosage, oral administration
- Hydrochlorothiazide (HCTZ): Encapsulated Hydrochlorothiazide 12.5 mg or 25 mg total daily dosage, oral administration with concomitant treatment consisting of lisinopril 10 mg total daily dosage, oral administration or losartan 50 mg total daily dosage, oral administration.
- Placebo: Placebo with concomitant treatment consisting of lisinopril 10 mg total daily dosage, oral administration or losartan 50 mg total daily dosage, oral administration.
Period: Overall Study
Arm/Group | Nebivolol | Hydrochlorothiazide (HCTZ) | Placebo
Started | 223 | 212 | 102
Completed | 178 | 174 | 90
Not Completed | 45 | 38 | 12
Not completed — Adverse Event | 23 | 14 | 2
Not completed — Lack of Efficacy | 2 | 2 | 2
Not completed — Protocol Violation | 6 | 9 | 1
Not completed — Withdrawal by Subject | 7 | 4 | 1
Not completed — Lost to Follow-up | 6 | 6 | 5
Not completed — Sponsor Terminated due to PI oversight | 0 | 1 | 0
Not completed — Poor compliance | 1 | 0 | 0
Not completed — Participated in two Nebivolol studies | 0 | 0 | 1
Not completed — Unconfirmed pregnancy | 0 | 1 | 0
Not completed — Randomization criteria not met | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Hydrochlorothiazide (HCTZ) | Placebo | Total
Number analyzed (Participants) | 223 | 212 | 102 | 537
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (9.6) | 55.7 (10.4) | 55.2 (11.3) | 55.1 (10.3)
Age, Customized [Count of Participants; unit: Participants]
  Patients 18 to 65 years of age | 190 | 172 | 81 | 443
  Patients greater than or equal to 65 years of age. | 33 | 40 | 21 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 97 | 38 | 236
  Male | 122 | 115 | 64 | 301
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 223 | 212 | 102 | 537

OUTCOME MEASURES:

1. Primary Outcome: Trough Seated Diastolic Blood Pressure
Description: Change from Baseline in Mean Seated Trough Cuff Diastolic Blood Pressure (DBP) at Week 12, Last Observation Carried Forward (LOCF).
Time Frame: Change from Baseline Visit 4 (Week 0) To Visit 8 (Week 12)
Population: The between-treatment-group comparison was performed by means of an analysis-of-covariance model with treatment group and study center as factors and baseline value as a covariate based on Intent-to-Treat (ITT) population. As pre-specified in the protocol, the change in seated DBP was performed between the nebivolol and placebo group.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 217 | 100
mm Hg | -9.4 (8.9) | -5.0 (9.5)

2. Secondary Outcome: Plasma Glucose Level After an Oral Glucose Tolerance Test
Description: Change from Baseline in Plasma Glucose 2 Hours Post-oral Glucose 75 grams, given as part of an Oral Glucose Tolerance Test (OGTT). Last Observation Carried Forward.
Time Frame: Change from Baseline Visit 3 or 4 (Week -2 or 0) To Visit 8 (Week 12)
Population: The between-treatment-group comparison was performed by means of an analysis-of-covariance model with treatment group and study center as factors and baseline value as a covariate based on Intent-to-Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: g/mL
Arm/Group | Nebivolol | Hydrochlorothiazide (HCTZ) | Placebo
Number analyzed (Participants) | 217 | 209 | 100
g/mL | 0.20 (0.190) | 0.31 (0.184) | -0.21 (0.247)

ADVERSE EVENTS:
Arm/Group | Nebivolol | Hydrochlorothiazide (HCTZ) | Placebo
Serious Adverse Events (participants affected / at risk) | 5/223 | 6/212 | 2/102
Other Adverse Events (participants affected / at risk) | 35/223 | 21/212 | 14/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=223) | Hydrochlorothiazide (HCTZ) (N=212) | Placebo (N=102)
Basal ganglia haemorrage (Nervous system disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Myocardial infaction (Cardiac disorders) | 0 | 2 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=223) | Hydrochlorothiazide (HCTZ) (N=212) | Placebo (N=102)
Bradycardia (Cardiac disorders) | 12 | 0 | 0
Headache (Nervous system disorders) | 12 | 12 | 7
Upper respiratory tract infection (Infections and infestations) | 12 | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute.